CLINICAL TRIAL: NCT02422381
Title: A Phase I/II Study of MK-3475 With Gemcitabine in Patients With Previously-Treated Advanced Non-small Cell Lung Cancer (NSCLC)
Brief Title: MK-3475 and Gemcitabine in Non-Small Cell Lung Cancer (NSCLC)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Providence Health & Services (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Providence Cancer Center, Earle A. Chiles Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-011A
Record Dates: First submitted 2015-03-20; First posted 2015-04-21 (Estimated); Results first posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: NSCLC; lung cancer; Gemzar; Pembrolizumab; Anti-PD-1; Immunotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — pembrolizumab; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MK-3475 + Gemcitabine (Experimental): 200mg MK-3475 200 given by IV infusion every 3 weeks, for 2 years, or until disease progression and Gemcitabine 1250 mg/m2 iv Days 1, 8 every 3 weeks, for maximum 6 cycles.
  Interventions: Drug: MK-3475; Drug: Gemcitabine

INTERVENTIONS:
Drug: MK-3475 — Investigational drug.
  Other Names: Anti-PD-1, Pembrolizumab
Drug: Gemcitabine — Standard care drug.
  Other Names: Gemzar

SUMMARY:
This is a study for patients with previously-treated advanced non-small cell lung cancer (NSCLC). The study will evaluate the safety of adding an investigational drug, MK-3475 to standard treatment with gemcitabine. The study will also try to identify the best dose of MK-3475 to give in combination with gemcitabine.

DETAILED DESCRIPTION:
This study is an open-label, non-randomized phase I study, followed by open-label non-randomized phase II study. The first cohort of patients will receive 200 milligrams (mg) of MK-3475 by intravenous infusion over a 21-day period called a cycle along with Gemcitabine 1250 mg/m2 given on Days 1 and 8 of each 21-day cycle for up to 6 cycles. Patients will be seen in the study clinic 12 times over 126 days for an evaluation of signs and symptoms that may represent drug toxicity. Patients may continue to receive MK-3475 (without gemcitabine) for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Women or men with advanced, histologically proven NSCLC.
* Patients must have received at least one but no more than three prior systemic therapies for advanced disease.
* Any toxicity related to prior therapies that, in the opinion of the investigator, would potentially be worsened with anti-PD1 therapy or gemcitabine should be resolved to less than Grade 1.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* Women of childbearing potential must have a negative pregnancy test
* Ability to give informed consent and comply with the protocol.
* Anticipated survival minimum 3 months.
* Prior therapy with investigational agents must have been completed at least 3 weeks prior to study enrollment.
* Patients must have normal organ and marrow function as seen on protocol-defined blood test results
* Archived tumor tissue (minimum of 8 slides for paraffin-embedded tumor tissue) available
* Measurable disease by RECIST 1.1 criteria.
* Treated brain metastases will be allowed, provided they are asymptomatic.
* Radiation for symptomatic lesions outside the Central nervous system (CNS) must have been completed at least 2 weeks prior to study enrollment.

Exclusion Criteria:

* Prior therapy with any anti-PD-1, anti-PD-L1, or anti-CTLA4 antibody.
* Prior therapy with gemcitabine.
* Prior complications from radiation, such as history of radiation pneumonitis or pulmonary edema that, in the opinion of the investigator, may have risk of increasing toxicity with anti-PD1 therapy.
* Active autoimmune disease except vitiligo or stable hypothyroidism.
* Active and ongoing steroid use, except for non-systemically absorbed treatments (such as inhaled or topical steroid therapy for asthma, cardiopulmonary disease (COPD), allergic rhinitis).
* Active other malignancy, except for controlled basal cell skin carcinoma.
* HIV positive and/or Hepatitis B or C positive.
* Other medical or psychiatric conditions that in the opinion of the Principal Investigator would preclude safe participation in this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-07-20 (Actual); Primary Completion 2019-01-09 (Actual); Study Completion 2026-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Sanborn, MD, Principal Investigator — Providence Health & Services
Locations (2):
- United States (2):
  - Providence Oncology & Hematology Care Clinic - Eastside, Portland, Oregon
  - Providence Oncology & Hematology Care Clinic - Westside, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Providence Cancer Center — http://oregon.providence.org/our-services/p/providence-cancer-center/

RESULTS

PARTICIPANT FLOW:
Groups:
- MK-3475 + Gemcitabine: 200mg MK-3475 200 given by IV infusion every 3 weeks, for 2 years, or until disease progression and Gemcitabine 1250 mg/m2 iv Days 1, 8 every 3 weeks, for maximum 6 cycles.
  MK-3475: Investigational drug.
  Gemcitabine: Standard care drug.
  Patients enrolled in the phase I and II portions were evaluated together for outcomes. There were no DLTs, so there was no dose de-escalation triggered and all 16 patients then received the same therapy, per protocol.
Period: Overall Study
Arm/Group | MK-3475 + Gemcitabine
Started | 16
Completed | 2
Not Completed | 14
Not completed — Death | 14

BASELINE CHARACTERISTICS:
Arm/Group | MK-3475 + Gemcitabine
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 11
Age, Continuous [Median (Full Range); unit: years] | 76 [60 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 16
Baseline ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) is a measure of functional status from scores ranging from 0 to 5. Baseline measure ECOG PS was collected during the screening physical exam. Lower scores indicated better outcomes.
  Participants
    ECOG PS 0 (Asymptomatic) | 2
    ECOG PS 1 (Symptomatic but completely ambulatory) | 14
    ECOG PS 2 (Symptomatic, <50% in bed during the day) | 0
    ECOG PS 3 (Symptomatic, >50% in bed, but not bedbound) | 0
    ECOG PS 4 (Bedbound) | 0
    ECOG PS 5 (Death) | 0
Tumor Histology [Count of Participants; unit: Participants]
  Adenocarcinoma | 12
  Squamous Cell Carcinoma | 1
  Non-Small Cell Lung Cancer (not otherwise specified) | 3

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicities
Description: Patients are seen in clinic 12 times over 126 days to determine any changes in signs or symptoms that may represent drug toxicity. Drug toxicity is defined as events that required holding or delaying treatment.
Time Frame: 126 Days (six 21-day cycles)
Measure: Count of Participants; unit: Participants
Arm/Group | MK-3475 + Gemcitabine
Number analyzed (Participants) | 16
Participants | 0

2. Secondary Outcome: Progression Free Survival
Description: Patients will have CT scans after every two cycles for up to 2 years to assess changes in tumor sizes.
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | MK-3475 + Gemcitabine
Number analyzed (Participants) | 16
months | 3.10 [2.60 to 5.68]

3. Secondary Outcome: Overall Survival
Description: Patients will be contacted every 12 weeks following end of treatment to determine survival status until death, withdrawal of consent, or the end of the study, whichever occurs first.
Time Frame: Every 12 weeks (up to 2 years)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | MK-3475 + Gemcitabine
Number analyzed (Participants) | 16
months | 8.20 [5.03 to 28.29]

4. Secondary Outcome: Disease Response
Description: Patients will have CT scans to assess changes in tumor sizes.
Time Frame: up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | MK-3475 + Gemcitabine
Number analyzed (Participants) | 16
Participants
  Complete Response | 0
  Partial Response | 2
  Stable Disease | 9
  Progressive Disease | 5

ADVERSE EVENTS:
Time Frame: Adverse events were collected over 6 21-day cycles (126 days). All-cause mortality was assessed up to 2 years from the end of treatment.
Arm/Group | MK-3475 + Gemcitabine
All-Cause Mortality (participants affected / at risk) | 14/16
Serious Adverse Events (participants affected / at risk) | 9/16
Other Adverse Events (participants affected / at risk) | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-3475 + Gemcitabine (N=16)
Acute hypoxemia respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Bowel obstruction (Gastrointestinal disorders) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 1 (1)
Dyspneic episode (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Fever (General disorders) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Transminitis (Hepatobiliary disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-3475 + Gemcitabine (N=16)
Abdominal bloating (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (5)
Abdominal soreness (Gastrointestinal disorders) | 1 (1)
Abdominal swelling (Gastrointestinal disorders) | 1 (1)
Absolute neutrophil count decreased (Investigations) | 2 (4)
Agitation (Psychiatric disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Alveolar hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 8 (9)
Anorexia (Metabolism and nutrition disorders) | 8 (9)
Anxiety (Psychiatric disorders) | 4 (4)
Arthralgias (Musculoskeletal and connective tissue disorders) | 2 (3)
Ascites (Gastrointestinal disorders) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Anosmia (Nervous system disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Bilateral leg edema (General disorders) | 1 (1)
Bilateral lower extremity edema (General disorders) | 1 (1)
Bilateral rhonchi (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Body aches (General disorders) | 2 (2)
Bronchitis (Infections and infestations) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Cancer pain (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 6 (7)
Cardiac chest pain (Cardiac disorders) | 1 (1)
Chest tightness (Cardiac disorders) | 2 (2)
Chills (General disorders) | 4 (4)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Coccyx pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cognitive changes (Nervous system disorders) | 1 (1)
Congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 8 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Creatinine increased (Investigations) | 4 (5)
Decreased breaths sounds (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 2 (3)
Depression (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 5 (5)
Dizziness (Nervous system disorders) | 1 (1)
Dog bite (Injury, poisoning and procedural complications) | 1 (1)
Dry cough (General disorders) | 1 (1)
Dry eyes (Eye disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dry oral mucosa (Gastrointestinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 (12)
Dysphagia (Gastrointestinal disorders) | 4 (4)
Dysruia (Renal and urinary disorders) | 1 (1)
Edema (General disorders) | 5 (7)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)
Excess sweating (Skin and subcutaneous tissue disorders) | 1 (1)
Fatigue (General disorders) | 13 (20)
Fever (General disorders) | 4 (6)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Flu like symptoms (General disorders) | 6 (7)
Frontal lobe burning sensation (Nervous system disorders) | 1 (1)
Paraesophageal hernia (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (3)
Hematuria (Renal and urinary disorders) | 2 (3)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hyperchloremic acidosis (Blood and lymphatic system disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 9 (9)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 3 (3)
Hypertension (Vascular disorders) | 3 (3)
Hyperuricemia (Metabolism and nutrition disorders) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 4 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 5 (5)
Hyponatremia (Metabolism and nutrition disorders) | 6 (7)
Hypophosphatemia (Metabolism and nutrition disorders) | 4 (4)
Hypotension (Vascular disorders) | 4 (4)
Hypouricemia (Blood and lymphatic system disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Ileal obstruction (Gastrointestinal disorders) | 1 (1)
Increasing pain (General disorders) | 1 (1)
Increasing productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1)
Insomnia (Psychiatric disorders) | 4 (4)
Left axillary pain (General disorders) | 1 (1)
Left hand infection (Infections and infestations) | 1 (1)
Left hip pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Left leg pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Left upper quadrant pain (General disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (2)
Malaise (General disorders) | 2 (2)
Mild Blurry Vision (Eye disorders) | 1 (1)
Muscle spasm (Musculoskeletal and connective tissue disorders) | 2 (3)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (6)
Nausea (Gastrointestinal disorders) | 12 (15)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neuropathy (Nervous system disorders) | 4 (4)
Neutrophil count decreased (Investigations) | 6 (6)
Oral lesions (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Oral thrush (Infections and infestations) | 1 (2)
Pain (General disorders) | 2 (2)
Pain in left flank (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain when swallowing (Gastrointestinal disorders) | 1 (1)
Paroxysmal atrial fibrillation episode (Cardiac disorders) | 1 (1)
Platelet count decreased (Investigations) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonia (Infections and infestations) | 3 (3)
Port discomfort (General disorders) | 1 (1)
Port site tenderness (General disorders) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 6 (8)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (7)
Rash (Skin and subcutaneous tissue disorders) | 3 (4)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1)
Rhonchi, right lung (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Right knee pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Right lateral thigh pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Right shoulder pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Right side lower neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Scrotal pain (Reproductive system and breast disorders) | 1 (1)
Sensitive skin (Skin and subcutaneous tissue disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Side pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 4 (4)
Skin breakdown around port site (General disorders) | 1 (1)
Cold sore (Infections and infestations) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Soreness at surgical incision (General disorders) | 1 (1)
Subcutaneous nodules in left upper arm (General disorders) | 1 (1)
Submandibular adenopathy (Infections and infestations) | 1 (1)
Swelling in ankle (Musculoskeletal and connective tissue disorders) | 1 (1)
Tender nodule on left upper foot (General disorders) | 1 (1)
Throat pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tingling in legs (Nervous system disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 2 (3)
Urinary retention (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
Vomiting (Gastrointestinal disorders) | 6 (8)
Weight loss (Investigations) | 2 (3)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 5 (8)
White blood cell decreased (Investigations) | 3 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-28): https://cdn.clinicaltrials.gov/large-docs/81/NCT02422381/Prot_SAP_000.pdf